CLINICAL TRIAL: NCT02594280
Title: Observational/Prospective Study for Benchmarking the Management of Glaucoma With Selective Laser Trabeculoplasty (SLT) or Trabecular Stent Bypass Microsurgery, Using the Diopsys Visual Evoked Potential/Pattern ERG Protocols
Brief Title: Benchmarking Management of Glaucoma Using the Diopsys VEP/PERG Protocols.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Diopsys, Inc. (Industry)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-UPMC-01; NCT02555436 (obsolete NCT alias)
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Selective Laser Trabeculoplasty (SLT)SLT: Monitor glaucoma patients that are scheduled to be treated with Selective Laser Trabeculoplasty (SLT) with VEP/PERG. The treatment is not dependent on the study.
- Trabecular stent bypass microsurgery: Monitor glaucoma patients that are scheduled to be treated with trabecular stent bypass microsurgery with VEP/PERG.The treatment is not dependent on the study.

SUMMARY:
Establish electrophysiological benchmarks, using the Diopsys Visual Evoked Potential/ Pattern ERG (VEP/PERG) protocols of populations with Glaucoma following: 1) Baseline VEP/ERG prior to treatment; and 2) VEP/PERG after treatment.

DETAILED DESCRIPTION:
The VEP and PERG have been proven and accepted as a viable clinical tool in the assessment of diseases of the retina ganglion cells. The Diopsys® Neuro Optic Vision Assessment Vision (NOVA) Testing System generates a battery of retinal responses evoked by viewing horizontal/checkerboard grating patterns with optimized contrast levels and visual field sizes.

Electrophysiological tests evaluate the function of the different structures constituting the visual nervous pathways (retina, optic nerve, optic tract, and chiasm, radiation and cerebral cortex). Among the various electrophysiological examinations, two very important tests are Electroretinograms (ERGs), which study the various retinal components, and Visual Evoked Potentials (VEPs) which study the visual pathway. These tests provide objective information on the function of the visual system even in those cases in which opacities of dioptric means (cataract, corneal leukoma) do not allow the direct observation of the retina and optic nerve, and may provide functional information in advance of structural changes.

Maculopathy and neuropathies are included in the long list of diseases of the visual pathway that permanently impair visual function. As there are considerable evidences related to the nature and evaluation of maculopathy and glaucomatous neuropathy, objective and reliable techniques are needed for visual function evaluation. By using PERG recordings, doctors are able to differentiate between normal subjects and subjects with ocular hypertension notwithstanding a normal optic disc and VF. PERG can provide important diagnostic information regarding the functional integrity of the macula and ganglion cells.

Based on a longitudinal study from Bascom Palmer Eye, abnormal retina function was recorded by PERG eight years before structural damage to the RNFL was detected. The study suggests that for glaucoma suspects it takes two years for a 10% change in PERG amplitude while it takes ten years for 10% change in RNFL.

The Diopsys® NOVA-pERG is a retinal biopotential that is evoked when a temporally phase-reversed horizontal/checkerboard grating pattern of constant total luminance is viewed. The contrast and viewing angle of the stimulus is optimized to elicit detection of dysfunction of the macula or the retinal ganglion cells selectively. The two NOVA-PERG reporting protocols are Contrast Sensitivity (CS) and Concentric Stimulus Fields (CSF). CS is optimized to detect dysfunctions of the retina that are sensitive to discrimination between different contrast levels while the CSF is optimized to localized pathologies in specific regions of the retina such as central vision and macula. Currently both protocols utilize steady-state technology.

The advantage of the Diopsys ERG as compared to traditional PERG is that it is non-invasive electrodes are attached to the eyelid and not the conjunctiva, and takes ten minutes to perform instead of 45. Patients do not been to be dark-adapted.

VEPs will be generated using a commercially available Diopsys NOVA System utilizing a fixed protocol. The stimulus will be presented on a 17-inch LCD monitor, running at 75 frames/s. Commercially available skin preparation and EEG paste will be used for recording of the SD-tVEP. Synchronized single-channel VEPs will be recorded, generating a time series of 1024 data points per analysis window. The room luminance will be maintained at scotopic conditions (<0.3 NITS). Preadaptation will be unnecessary for the SD-tVEP recordings. Multiple tests are run to comprise one SD-tVEP protocol. One complete NOVA-VEP (FP) presents a stimulus for a maximum of 1 minute and 46 seconds.

In all cases, the display will be viewed through natural pupils (undilated) with optimal refractive correction in place. The viewing distance will be set to 1 m, yielding a total display viewing angle of 15.5 degrees. The square black/white checkerboard pattern reversal stimulus has a height and width of 27 cm with a red circular ring used as a fixation target. The diameter of the target is approximately 1.5 cm with a ring thickness of 1.5 mm. The target ring will be centered on the stimulus. The check size will be 29.0 minutes of arc. Two pattern contrasts will be used in the study, based on earlier studies that suggested that differential contrast stimulation could affect the NOVA-VEP (FP) waveforms. The first pattern will have a Michelson contrast of 15%. The second pattern will have a Michelson contrast of 85%. These two patterns are referred to as LC (Low contrast) and HC (High contrast) respectively.

During a recording session, the contrast polarity of each stimulus check will be temporally modulated at a reversal frequency of 1 Hz (2 pattern reversals equates to 1 reversal cycle); therefore, each reversal occurs at 2 Hz or twice per second. This stimulus is termed a pattern reversal stimulus and has a duty cycle of 50%. The 15% and 85% contrast stimuli will be presented for each eye (the fellow eye was covered) for 15 seconds. The right eye will be the first one to be tested for all patients.

In preparation for recording, the skin at each electrode site will be scrubbed with Nuprep using a cotton gauze pad. Electrodes will be fixed in position with Ten20 conductive paste and secured with a small gauze pad with conductive paste applied. Electrode impedance will be maintained below 10 kohm and typically kept below 5 kohm.

The Pattern Electroretinogram (PERG) will be recorded using a commercially available system Diopsys® NOVA (Diopsys, Inc. Pine Brook, New Jersey). The testing protocol will include the Concentric Stimulus Field (CSF).

Subjects will be fitted with the appropriate correction for a viewing distance of 24 inches and will be instructed to fixate on a target at the center of stimulus monitor. The test will be performed in a dark room to standardized environment luminance, free of visual and audible distractions. The subject will be comfortable seated facing the stimulus monitor. The patient's seated height will be adjusted so the eye stays in a horizontal plane with the center of the monitor. The test will be performed without pupil dilation and subjects will be allowed to blink freely.

The PERG will be recorded from the study eye by means of hypoallergenic skin sensors Silver/Silver Chloride ink (Diopsys® proprietary Skin Sensor) on the lower eyelids. The reference sensor will be located in the contralateral eyelid and ground sensor in the central forehead area (Fz). The skin will be prepared by cleaning with eyelid cleanser (OCuSOFT®) to ensure good and stable electrical conductivity, keeping the impedances bellow 5 kohm.

The stimulus will be presented on a gamma corrected Acer V173BM 17-inch LCD monitor, having a refresh rate of 75 frames / second. The CSF pattern stimulus will consist of black/white horizontal gratings (24° and 16° circular field, 98% contrast and 102.28 candelas/m2 mean luminance), reversing at 15 reversals/second) with a duration of 25 seconds. A red spinning ring will be used as a fixation target with a diameter of 1 cm and 1 mm of thickness. This target ring will be at the corner of four checks, centered on the stimulus field.

A test will be categorized as non-reliable if Phase Variance is greater than 0.4 and/or if the Magnitude Variance to Magnitude Ratio (VMR) is greater than 2.9 and/or if more than 4 artifacts are detected. The FERG test results will be saved in an SQL database and presented in a report form to be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient will have repeatable abnormal SAP results (pattern standard deviation with p ≤5% and/or Glaucoma Hemifield Test outside normal limits)
* Glaucomatous optic disc appearance (those with cup to disc area ratio, rim thinning or RNFL defects indicative of glaucoma)
* Repeatable intraocular pressure ≥23 mmHg, in at least one eye.
* The last SAP test of all participants will be classified following the Glaucoma Staying System (GSS).

Exclusion Criteria:

* A spherical refraction outside + 5.0 D and cylinder correction outside + 3.0 D.
* Intraocular surgery in the study eye (except non-complicated cataract or refractive surgery performed less than 1 year before enrollment).
* Any prior vitrectomy
* Any prior macular or pan retinal photocoagulation laser
* History of neurologic condition known to affect visual function.
* Inability to obtain a reliable PERG/VEP test.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is a group of glaucoma patients that are scheduled for 1) Selective Laser Trabeculoplasty or 2) Trabecular stent bypass microsurgery as a treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-02-15 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
VEP Amplitude at 15% Contrast | Within 1 month prior to treatment
  Record the VEP Amplitude at 15% contrast stimulus.
VEP Amplitude at 15% Contrast | 3 months post treatment
  Record the VEP Amplitude at 15% contrast stimulus.
VEP Amplitude at 15% Contrast | 6 months post treatment
  Record the VEP Amplitude at 15% contrast stimulus
VEP Latency at 15% Contrast | Within 1 month prior to treatment
  Record the VEP Latency at 15% contrast stimulus.
VEP Latency at 15% Contrast | 3 months post treatment
  Record the VEP Latency at 15% contrast stimulus
VEP Latency at 15% Contrast | 6 months post treatment
  Record the VEP Latency at 15% contrast stimulus
VEP Amplitude at 85% Contrast | Within 1 month prior to treatment
  Record the VEP Amplitude at 85% contrast stimulus.
VEP Amplitude at 85% Contrast | 3 months post treatment
  Record the VEP Amplitude at 85% contrast stimulus.
VEP Amplitude at 85% Contrast | 6 months post treatment
  Record the VEP Amplitude at 85% contrast stimulus.
VEP Latency at 85% Contrast | Within 1 month prior to treatment
  Record the VEP Latency at 85% contrast stimulus
VEP Latency at 85% Contrast | 3 months post treatment
  Record the VEP Latency at 85% contrast stimulus
VEP Latency at 85% Contrast | 6 months post treatment
  Record the VEP Latency at 85% contrast stimulus
PERG Magnitude at 16 degree stimulus | Within 1 month prior to treatment
  Record the PERG Magnitude at 16 degree stimulus
PERG Magnitude at 16 degree stimulus | 3 months post treatment
  Record the PERG Magnitude at 16 degree stimulus
PERG Magnitude at 16 degree stimulus | 6 months post treatment
  Record the PERG Magnitude at 16 degree stimulus
PERG MagnitudeD at 16 degree stimulus | Within 1 month prior to treatment
  Record the PERG MagnitudeD at 16 degree stimulus
PERG MagnitudeD at 16 degree stimulus | 3 months post treatment
  Record the PERG MagnitudeD at 16 degree stimulus
PERG MagnitudeD at 16 degree stimulus | 6 months post treatment
  Record the PERG MagnitudeD at 16 degree stimulus
PERG Magnitude at 24 degree stimulus | Within 1 month prior to treatment
  Record the PERG Magnitude at 24 degree stimulus
PERG Magnitude at 24 degree stimulus | 3 months post treatment
  Record the PERG Magnitude at 24 degree stimulus
PERG Magnitude at 24 degree stimulus | 6 months post treatment
  Record the PERG Magnitude at 24 degree stimulus
PERG MagnitudeD at 24 degree stimulus | Within 1 month prior to treatment
  Record the PERG MagnitudeD at 24 degree stimulus
PERG MagnitudeD at 24 degree stimulus | 3 months post treatment
  Record the PERG MagnitudeD at 24 degree stimulus
PERG MagnitudeD at 24 degree stimulus | 6 months post treatment
  Record the PERG MagnitudeD at 24 degree stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Wollstein Gadi, MD, Principal Investigator — University of Pittsburgh

REFERENCES:
- [Background] Bach M, Brigell MG, Hawlina M, Holder GE, Johnson MA, McCulloch DL, Meigen T, Viswanathan S. ISCEV standard for clinical pattern electroretinography (PERG): 2012 update. Doc Ophthalmol. 2013 Feb;126(1):1-7. doi: 10.1007/s10633-012-9353-y. Epub 2012 Oct 17. PMID 23073702
- [Background] Banitt MR, Ventura LM, Feuer WJ, Savatovsky E, Luna G, Shif O, Bosse B, Porciatti V. Progressive loss of retinal ganglion cell function precedes structural loss by several years in glaucoma suspects. Invest Ophthalmol Vis Sci. 2013 Mar 28;54(3):2346-52. doi: 10.1167/iovs.12-11026. PMID 23412088
- [Background] Bode SF, Jehle T, Bach M. Pattern electroretinogram in glaucoma suspects: new findings from a longitudinal study. Invest Ophthalmol Vis Sci. 2011 Jun 16;52(7):4300-6. doi: 10.1167/iovs.10-6381. PMID 21372021
- [Background] Parisi V, Miglior S, Manni G, Centofanti M, Bucci MG. Clinical ability of pattern electroretinograms and visual evoked potentials in detecting visual dysfunction in ocular hypertension and glaucoma. Ophthalmology. 2006 Feb;113(2):216-28. doi: 10.1016/j.ophtha.2005.10.044. Epub 2006 Jan 10. PMID 16406535
- [Background] Dodt E. The electrical response of the human eye to patterned stimuli: clinical observations. Doc Ophthalmol. 1987 Mar;65(3):271-86. doi: 10.1007/BF00149934. PMID 3678000
- [Background] Carr MD RE. The Pattern Electroretinogram (PERG). Paper presented at: NANOS, 1988.
- [Background] Ventura LM, Porciatti V. Pattern electroretinogram in glaucoma. Curr Opin Ophthalmol. 2006 Apr;17(2):196-202. doi: 10.1097/01.icu.0000193082.44938.3c. PMID 16552256
- [Background] Bach M, Unsoeld AS, Philippin H, Staubach F, Maier P, Walter HS, Bomer TG, Funk J. Pattern ERG as an early glaucoma indicator in ocular hypertension: a long-term, prospective study. Invest Ophthalmol Vis Sci. 2006 Nov;47(11):4881-7. doi: 10.1167/iovs.05-0875. PMID 17065502
- [Background] Kono Y, Jonas JB, Zangwill L, Berry CC, Weinreb RN. Agreement of measurement of parapapillary atrophy with confocal scanning laser ophthalmoscopy and planimetry of photographs. J Glaucoma. 1999 Apr;8(2):105-10. PMID 10209726
- [Background] Holder GE. Pattern electroretinography (PERG) and an integrated approach to visual pathway diagnosis. Prog Retin Eye Res. 2001 Jul;20(4):531-61. doi: 10.1016/s1350-9462(00)00030-6. PMID 11390258